CLINICAL TRIAL: NCT01262924
Title: A Phase III, Blinded, Randomised, Monocentre, Comparative Clinical Study of the Immunogenicity, Reactogenicity and Safety of a Single Booster Dose of SB Biologicals' Candidate dTpa and pa Vaccines and SB Biologicals' Licensed Td Vaccine in Healthy Adults Aged ≥18 Years
Brief Title: Study of Reduced-antigen-content Acellular Pertussis Vaccine and Diphtheria-Tetanus-Acellular Pertussis Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 263855/003
Record Dates: First submitted 2010-12-16; First posted 2010-12-17 (Estimated); Last update posted 2010-12-17 (Estimated); Status verified 2010-12

CONDITIONS: Diphteria, Tetanus and Pertussis
Keywords: Booster vaccination
MeSH Terms: conditions — Tetanus; Whooping Cough

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Group A (Experimental): dTPa vaccine
  Interventions: Biological: GSK Biologicals' reduced-antigen-content diphtheria-tetanus-acellular pertussis vaccine
- Group B (Experimental): Pa vaccine
  Interventions: Biological: GSK Biologicals' reduced-antigen-content acellular pertussis vaccine
- Group C (Active Comparator): Tedivax-Adult™/ Td-Rix™
  Interventions: Biological: Tedivax-Adult™/ Td-Rix™

INTERVENTIONS:
Biological: GSK Biologicals' reduced-antigen-content diphtheria-tetanus-acellular pertussis vaccine — Intramuscular, single dose
  Arms: Group A
Biological: GSK Biologicals' reduced-antigen-content acellular pertussis vaccine — Intramuscular, single dose
  Arms: Group B
Biological: Tedivax-Adult™/ Td-Rix™ — Intramuscular, single dose or 2 doses (in the annex phase)
  Arms: Group C

SUMMARY:
The purpose of this study is to assess the immunogenicity and reactogenicity of GlaxoSmithKline (GSK) Biologicals' (formerly, SmithKline Beecham Biologicals) reduced-antigen-content acellular pertussis vaccine and reduced-antigen-content diphtheria-tetanus-acellular pertussis vaccine in comparison with Tedivax-Adult™/ Td-Rix™

ELIGIBILITY:
Inclusion Criteria:

* A male or female aged ≥18 years at the time of vaccination
* Free of obvious health problems as established by medical history and clinical examination before entering into the study
* Written informed consent obtained from the subject
* If the subject is female, she must be of non-childbearing potential , i.e., either surgically sterilised or one year post-menopausal; or, if of childbearing potential, she must be abstinent or have used adequate contraceptive precautions for 30 days prior to vaccination, have a negative pregnancy test and must agree to continue such precautions for two months after completion of the vaccination series.

For the annex phase of this study, subjects must meet the inclusion criteria mentioned above. In addition, subjects must have received either reduced-antigen-content diphtheria-tetanus or diphtheria-tetanus-acellular pertussis vaccine in the initial phase of the study and not responded to either the diphtheria or tetanus toxoid..

Exclusion Criteria:

* Vaccination against diphtheria and/or tetanus within the previous five years
* Vaccination against pertussis since childhood
* History of diphtheria and/or tetanus
* Known history of pertussis within the previous five years
* Known exposure to diphtheria or pertussis within the previous five years
* Known history of non-response to diphtheria, tetanus or pertussis vaccine
* Use of any investigational or non-registered drug or vaccine other than the study vaccine(s) during the study period or within 30 days/ 5 half-lives preceding the dose of study vaccine
* Administration of chronic immunosuppressants or other immune-modifying drugs within six months/ 5 half-lives of vaccination.
* Planned administration/ administration of a vaccine not foreseen by the study protocol during the period starting from 30 days before vaccination and ending 30 days after
* Administration of immunoglobulins and/or any blood products within the three months preceding vaccination or planned administration/ administration during the study period
* Any confirmed or suspected immunosuppressive or immunodeficient condition
* Pregnant or lactating female
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine
* Hypersensitivity to any component of the vaccines
* Acute disease at the time of enrolment
* Oral temperature of ≥37.5°C (99.5°F)
* Any of the following having occurred after previous administration of diphtheria-tetanus-pertussis vaccine or diptheria and tetanus vaccines
* An immediate anaphylactic reaction
* Signs of encephalopathy
* Any of the following having occurred after previous administration of diphtheria-tetanus-pertussis vaccine alone or in combination with other antigens:
* Rectal temperature ≥40.5°C within 48 hours of vaccination and not due to another identifiable cause
* Collapse or shock-like state within 48 hours of vaccination
* Persistent, inconsolable screaming or crying lasting ≥3 hours within 48 hours of vaccination
* Convulsions with or without fever, occurring within 3 days of vaccination

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 1997-10; Primary Completion 1998-12 (Actual); Study Completion 1998-12 (Actual)

PRIMARY OUTCOMES:
Immunogenicity with respect to components of the study vaccines (in subjects receiving the dTpa vaccine and Tedivax-Adult™/ Td-Rix™) | One month after the booster dose (Month 1)

SECONDARY OUTCOMES:
Immunogenicity with respect to components of the study vaccines (in subjects receiving the dTpa, pa vaccines and Tedivax-Adult™/ Td-Rix™) | One month after the booster dose (Month 1)
Occurrence of solicited local adverse experiences | During the 15-day (Day 0-14) follow-up period after vaccination
Occurrence of solicited general adverse experiences | During the 15-day (Day 0-14) follow-up period after vaccination
Occurrence of unsolicited symptoms | Within the 31-day (Day 0 -30) follow-up period after vaccination
Occurrence of any serious adverse experiences | Within the 31-day (Day 0 -30) follow-up period after vaccination
Lymphoproliferation specific for pertussis toxoid, filamentous haemagglutinin and pertactin/ Cell mediated immunity response | At pre-vaccination (Day 0) and Month 1 post-vaccination
Immunogenicity with respect to components of the study vaccines (in subjects who did not respond to diphtheria or tetanus toxoid after the first booster dose) | One month after the second and third booster dose (Month 12)
Occurrence of solicited local adverse experiences (in subjects who did not respond to diphtheria or tetanus toxoid after the first booster dose) | During the 15-day (Day 0-14) follow-up period after the second and third vaccine dose
Occurrence of solicited general adverse experiences (in subjects who did not respond to diphtheria or tetanus toxoid after the first booster dose) | During the 15-day (Day 0-14) follow-up period after the second and third vaccine dose
Occurrenceof unsolicited symptoms (in subjects who did not respond to diphtheria or tetanus toxoid after the first booster dose) | Within the 31-day (Day 0 -30) follow-up period after vaccination after the second and third vaccine dose
Occurrence of any serious adverse experiences (in subjects who did not respond to diphtheria or tetanus toxoid after the first booster dose) | Within the 31-day (Day 0 -30) follow-up period after vaccination after the second and third vaccine dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Result] Van Damme P, Burgess M. Immunogenicity of a combined diphtheria-tetanus-acellular pertussis vaccine in adults. Vaccine. 2004 Jan 2;22(3-4):305-8. doi: 10.1016/j.vaccine.2003.08.012. PMID 14670310